CLINICAL TRIAL: NCT05112315
Title: Clinical Impact of the IBox As an Early Intervention TooL: a Prospective Randomised Controlled Trial to Assess the Use of a Software Predicting Allograft Survival in the Follow-up of Kidney Transplanted Patients.
Brief Title: Clinical Impact of the IBox As an Early Intervention TooL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Predict4Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TF-Form-124
Record Dates: First submitted 2021-10-19; First posted 2021-11-08 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Kidney Diseases; Kidney Disease, Chronic; Kidney Transplant Rejection; Kidney Transplant; Complications; Kidney Failure; Kidney Failure, Chronic; Kidney Dysfunction
Keywords: Chronic Kidney Disease; Kidney Transplant; IBox; Predigraft; Kidney allograft; Prediction; Rejection; Allograft survival
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency; Kidney Failure, Chronic; Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: randomized 1:1 , controlled, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Predigraft (Experimental): Subjects will have a clinical follow-up based on site standard of care and benefit from follow-up using Predigraft in addition of the standard of care: the investigator will receive an alert every time there is a subject's instability, instability based on the following criteria: allograft survival assessed by iBox decreased by at least 5% in the last 12 months.
  Interventions: Device: Predigraft
- Standard of Care (No Intervention): Subjects will have a clinical follow-up based on site standard of care.

INTERVENTIONS:
Device: Predigraft — The Subject randomized to the Predigraft will benefit from Predigraft, a remote monitoring software that issues an alert to the investigator when the allograft survival prediction calculated by the iBox algorithm is decreasing. This follow-up is on top of the site's standard of care.
  Other Names: Remote monitoring
  Arms: Predigraft

SUMMARY:
International, multicentre, randomized 1:1 controlled trial to prove the clinical and medico economic benefits of the medical device Predigraft, by showing that the use of Predigraft could improve patient's follow-up.

DETAILED DESCRIPTION:
The study aims to demonstrate improvement of the prevalence of biopsies leading to therapeutic change in the Predigraft group compared to the Standard of care group in kidney transplanted patients.

It is hypothesized that using Predigraft as a monitoring tool will help the physician detect earlier and more often abnormalities with the patient allograft. This should lead to an increased number of biopsies leading to therapeutic change. These biopsies should be performed earlier than without the iBox monitoring tool. This would improve long-term allograft function, kidney allograft and patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age ≥ 18 years old at the time of consent.
* Patients receiving a living or deceased donor kidney allograft.
* Patients transplanted at least 3 months before inclusion.
* Patients who signed the informed consent form and are willing to comply with study procedures.

Exclusion Criteria:

* Combined transplant (i.e. heart-kidney, liver-kidney).
* Patients who are unable or unwilling to comply with study procedures.
* Vulnerable patients (minors, protected adults, legally detained).
* Patients participating in other interventional studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
number of biopsies leading to therapeutic change | 18 months
  number of biopsies leading to therapeutic change by the end of the follow-up (18 months).

SECONDARY OUTCOMES:
Lapse of time between the detection of kidney allograft instability and the biospy | 18 months
  Lapse of time between the detection of kidney allograft instability (i.e. Predigraft alert on patient's instability) and performing the biopsy.
Renal function | 18 months
  Renal function estimated by eGFR
Patient outcome | 18 months
  Patient outcome evaluated by a composite endpoint: graft loss + patient death + eGFR < 30 mL/min/1.73m2 by the end of the follow-up.
iBox predicted allograft survival | 18 months
  iBox predicted allograft survival: 7-year kidney allograft predictions by the end of the follow-up.
Number of therapeutic changes | 18 months
  Number of therapeutic changes by the end of the follow-up.
Number of unnecessary biopsies | 18 months
  Number of unnecessary biopsies by the end of the follow-up.

OTHER OUTCOMES:
Patient related outcome measures | 18 months
  Patient related outcome measures: results of SF-36 (36-Item Short Form Health Survey) (quality of life: score 0 to 100 / 0 being the worst perception of health status) questionnaire at the end of the follow-up compared to baseline.
Medico-economic evaluation | 18 months
  Medico-economic evaluation based on days of hospitalization, treatment cost and return to dialysis at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre LOUPY, Pr, Study Chair — Necker Hospital, Paris, France; Carmen LEFAUCHEUR, Pr, Principal Investigator — St Louis Hospital, Paris, France
Locations (16):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- France (4):
  - Hôpital Saint-Louis, Paris, France
  - Hôpital Tenon, Paris, France
  - CHU Rangueil, Toulouse, France
  - Hôpital Necker, Paris
- Germany (2):
  - Universitätsklinikum Düsseldorf AÖR, Düsseldorf
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Sourasky Medical Center - Ichilov Hospital, Tel Aviv, Israel
- Spain (3):
  - Hospital Del Mar - Parc de Salut Mar, Barcelona
  - Fundació Puigvert, Barcelona
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (5):
  - Queen Elizabeth Hospital, Birmingham
  - Leeds Teaching Hospital NHS Trust, Leeds
  - Guy's & Saint Thomas' NHS Foundation Trust, London
  - King's College Hospital, London
  - Oxford Transplant Centre, Oxford

IPD SHARING:
Plan to Share IPD: No
Data will be communicated to other researchers in an aggregated manner